CLINICAL TRIAL: NCT04129918
Title: Effects of Light and Sound Modification on Sleep Quality and Circadian Rhythm in the Medical Intensive Care Unit Patients
Brief Title: Effects of Light and Sound Modification on Sleep Quality and Circadian Rhythm in the MICU Patients
Acronym: MICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20190804R
Record Dates: First submitted 2019-10-13; First posted 2019-10-17 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-01

CONDITIONS: Intensive Care Unit; Ventilator; Sleep Quality; Circadian Rhythm
Keywords: intensive care unit; sleep quality; circadian rhythm
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Light; Ear Protective Devices

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized control trial in the medical intensive care unit of the Shin Kong Wu Ho-Su Memorial Hospital.
Who Masked: Outcomes Assessor
Masking Description: The study was conducted on 126 patients with 56 subjects in experimental group and 56 in control group in the MICU. Effect of ear plugs & eye mask on sleep among ICU patients: a randomized control trial The participants were randomly divided into two groups: with ear plugs and eye mask (experimental group) for 3 successive nights and without ear plugs and eye mask (control group). participants were provided a Sequentially numbered opaque sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): ear plugs and eye mask for 3 successive nights
  Interventions: Behavioral: light and sound modification (earplugs and eye masks)
- control group (No Intervention): without ear plugs and eye mask

INTERVENTIONS:
Behavioral: light and sound modification (earplugs and eye masks) — In the experimental group，the patients used earplugs and eye masks during nighttime sleep.
  Arms: experimental group

SUMMARY:
This study will investigate the effectiveness of light and sound modification in improving sleep qualit , and circadian rhythms in MICU patients with Mechanical Ventilation in Taiwan.

Hypothesis:

1. The sleep quality in intervention group is significant improving than usual-care group at Day 1 (after the first intervention), Day 2 (after the second intervention), and Day 3 (after the third intervention).
2. The circadian rhythm in intervention group is significant improving than usual-care group at Day 1 (after the first intervention), Day 2 (after the second intervention), Day 3 (after the third intervention).

DETAILED DESCRIPTION:
The subjects were divided into experimental and control groups. And the improving quality of sleep intervention was provided only in experimental group. In the experimental group，the patients used earplugs and eye masks during nighttime sleep. In the control group, the received routine intensive care.

ELIGIBILITY:
Inclusion Criteria:

1. ICU stay for 7 days
2. Endotracheal or Tracheostomy patients

Exclusion Criteria:

1. Patients with ear injury
2. Hearing impairment
3. Eye disease or injuries

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Subjective sleep quality | baseline after recruited] using Chinese version of Richards-Campbell Sleep Questionnaire
  Subjective sleep quality
Subjective sleep quality | Day 1 after recruited] using Chinese version of Richards-Campbell Sleep Questionnaire
  Subjective sleep quality
Subjective sleep quality | Day 2 after recruited] using Chinese version of Richards-Campbell Sleep Questionnaire
  Subjective sleep quality
Subjective sleep quality | Day 3 after recruited] using Chinese version of Richards-Campbell Sleep Questionnaire
  Subjective sleep quality

SECONDARY OUTCOMES:
Objective sleep quality | baseline, Day 1, Day 2, and Day 3] using Actigraphy
  Objective sleep quality
Circadian rhythms | baseline, Day 1, Day 2, and Day 3] using Actigraphy
  Circadian rhythms including 24-h autocorrelation coefficient (r24), in bed less than out of bed dichotomy index (I<O) collection, Mesor, Amplitude, and Acrophase from actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Mei Chen, PhD, Study Chair — alice@ntunhs.edu.tw
Locations (1):
- ShinKongHospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
partial collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 12 months after publication
Access Criteria: Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).

REFERENCES:
- [Result] Pisani MA, Friese RS, Gehlbach BK, Schwab RJ, Weinhouse GL, Jones SF. Sleep in the intensive care unit. Am J Respir Crit Care Med. 2015 Apr 1;191(7):731-8. doi: 10.1164/rccm.201411-2099CI. PMID 25594808
- [Result] Kamdar BB, Niessen T, Colantuoni E, King LM, Neufeld KJ, Bienvenu OJ, Rowden AM, Collop NA, Needham DM. Delirium transitions in the medical ICU: exploring the role of sleep quality and other factors. Crit Care Med. 2015 Jan;43(1):135-141. doi: 10.1097/CCM.0000000000000610. PMID 25230376
- [Result] Boyko Y, Toft P, Ording H, Lauridsen JT, Nikolic M, Jennum P. Atypical sleep in critically ill patients on mechanical ventilation is associated with increased mortality. Sleep Breath. 2019 Mar;23(1):379-388. doi: 10.1007/s11325-018-1718-3. Epub 2018 Sep 13. PMID 30215172
- [Result] Delaney LJ, Currie MJ, Huang HC, Litton E, Wibrow B, Lopez V, Haren FV. Investigating the application of motion accelerometers as a sleep monitoring technique and the clinical burden of the intensive care environment on sleep quality: study protocol for a prospective observational study in Australia. BMJ Open. 2018 Jan 21;8(1):e019704. doi: 10.1136/bmjopen-2017-019704. PMID 29358448
- [Result] Solverson KJ, Easton PA, Doig CJ. Assessment of sleep quality post-hospital discharge in survivors of critical illness. Respir Med. 2016 May;114:97-102. doi: 10.1016/j.rmed.2016.03.009. Epub 2016 Mar 21. PMID 27109818
- [Result] Beltrami FG, Nguyen XL, Pichereau C, Maury E, Fleury B, Fagondes S. Sleep in the intensive care unit. J Bras Pneumol. 2015 Nov-Dec;41(6):539-46. doi: 10.1590/S1806-37562015000000056. PMID 26785964
- [Result] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Result] Horsten S, Reinke L, Absalom AR, Tulleken JE. Systematic review of the effects of intensive-care-unit noise on sleep of healthy subjects and the critically ill. Br J Anaesth. 2018 Mar;120(3):443-452. doi: 10.1016/j.bja.2017.09.006. Epub 2017 Nov 23. PMID 29452801